CLINICAL TRIAL: NCT02147717
Title: Laser Acupuncture and Pain Management in Preterm Infants Undergoing Patent Ductus Arteriosus Ligation
Acronym: ELAPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P 130602
Record Dates: First submitted 2014-05-19; First posted 2014-05-28 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2016-08

CONDITIONS: Preterm Newborns
Keywords: preterm newborns; Transfontanellar ultrafast doppler; Acupuncture; perioperative pain; surgery of the ductus arteriosus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser stimulation (Experimental): Laser stimulation plus opioid treatment before ETS. Low level laser acupuncture, 670 nm, 10Hz, 0,3 J per acupoint, 6 points per neonate (Zu san li, He Gu, Nei Guan) marquage CE, premio 30 laser duo de Sedatelec. Overall 3 minutes of treatment.
  This sequence will be repeated 4 times during the study (1 hour before surgery and every 12 hours after surgery)
  Interventions: Device: Laser stimulation
- fake laser stimulation (Placebo Comparator): newborns have the same preparation procedure as the intervention to put them under the same conditions group. The laser pen is turned off, off-voltage
  Interventions: Device: Fake laser stimulation

INTERVENTIONS:
Device: Laser stimulation — Infants will be divided in 2 groups:
  * Placebo group: Placebo (fake laser stimulation) plus opioid treatment before ETS
  * Experimental group: Laser stimulation plus opioid treatment before ETS. Low level laser acupuncture, 670 nm, 10Hz, 0,3 J per acupoint, 6 points per neonate (Zu san li, He Gu, Nei Guan) marquage CE, premio 30 laser duo de Sedatelec. Overall 3 minutes of treatment.
  This sequence will be repeated 4 times during the study (1 hour before surgery and every 12 hours after surgery)
  Arms: Laser stimulation
Device: Fake laser stimulation — newborns have the same preparation procedure as the intervention to put them under the same conditions group. The laser pen is turned off, off-voltage
  Arms: fake laser stimulation

SUMMARY:
Prospective study, controlled, randomized, single-center, blinded, which aims to evaluate the effect of laser acupuncture in the treatment of perioperative pain during tracheal suction after patent ductus arteriosus ligation in preterm infants.

DETAILED DESCRIPTION:
management of pain in preterm infants is essential because it is exposed to repetitive movements painful and invasive miners such as surgical treatment of the ductus arteriosus which is accompanied by respiratory instability, increased consumption analgesics. Acupuncture has shown its analgesic efficacy in numerous studies in children and adults. Acupuncture (laser) is a simple, fast method without side effect used in children, but no study exists on the effect of acupuncture in the treatment of perioperative pain in addition to pharmacologic agents in preterm infants. Hypothesis: acupuncture reduce pain and discomfort after surgery of the ductus arteriosus in preterm infants in addition to pharmacologic agents

Main objective:

Assessing the contribution of laser acupuncture on the pain management during endotracheal suctioning (ETS) after surgery ductus arteriosus in preterm infants

ELIGIBILITY:
Inclusion Criteria:

* Preterm infant born between 24 +0 and 32 +6 j GA
* Ductus arteriosus surgery scheduled in Robert Debré hospital
* Informed consent of the holders of the exercise of parental authority
* Child beneficiary of a social security scheme (excluding AME)

Exclusion Criteria:

* Obvious underlying disease (genetic, metabolic)

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Behavioral pain scale (COMFORT scale) | 48 hours post-operative
  Behavioral pain scale (COMFORT scale) studied at a painful procedure (endotracheal suctioning, ETS) with a regular assessment in perioperative. All the ETS will videotaped with a color digital camera by the research assistant.

SECONDARY OUTCOMES:
Behavioral pain scale (DAN scale and EDIN scale) | 48hours postoperative
  Behavioral pain scale during ETS (DAN scale) and after ETS (EDIN scale)
Consumption of morphine | 48 hours postoperative
  Consumption of morphine (cumulative mg / kg dose) from surgery to 48h postoperative
Measurement of FIO2 | 48 hours postoperative
  Measurement of FIO2, mode of mechanical ventilation after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Biran Valérie, PHD, Principal Investigator — APHP
Locations (1):
- Hôpital Robert Debré, Paris, France